CLINICAL TRIAL: NCT00981578
Title: A Feasibility Study to Evaluate the Safety and Initial Effectiveness of ExAblate MR Guided Focused Ultrasound Surgery in the Treatment of Pain Resulting From Metastatic Bone Tumors With the ExAblate 2100 Conformal Bone System
Brief Title: ExAblate Conformal Bone System Treatment of Metastatic Bone Tumors for the Palliation of Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to low enrollment.
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM010
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Bone Metastases
Keywords: bone cancer; pain palliation; metastasis; breast cancer; lung cancer; prostate cancer; cancer related pain; tumors
MeSH Terms: conditions — Bone Neoplasms; Neoplasm Metastasis; Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Cancer Pain; Neoplasms

ARMS (1):
- ExAblate 2100 Treatment (Experimental): ExAblate 2100 ablation for the treatment of painful bone metastases.
  Interventions: Device: ExAblate 2100

INTERVENTIONS:
Device: ExAblate 2100 — Conformal Bone System
  Other Names: Focused ultrasound ablation, MRgFUS

SUMMARY:
A study to evaluate the safety and initial effectiveness of the ExAblate 2100 Conformal Bone System in the treatment of pain resulting from metastatic bone tumors.

DETAILED DESCRIPTION:
Bone is the third most common organ involved by metastatic disease behind lung and liver [6]. In breast cancer, bone is the second most common site of metastatic spread, and 90% of patients dying of breast cancer have bone metastasis. Breast and prostate cancer metastasize to bone most frequently, which reflects the high incidence of both these tumors, as well as their prolonged clinical courses. Post-cancer survival has increased with improvement in early detection and treatments. As a consequence, the number of patients developing metastatic bone disease during their lifetime has also increased.

Current treatments for patients with bone metastases are primarily palliative and include localized therapies (radiation and surgery), systemic therapies (chemotherapy, hormonal therapy, radiopharmaceutical, and bisphosphonates although the primary goal of the use of these therapies are often to address the disease itself), and analgesics (opioids and non-steroidal anti-inflammatory drugs). Recently, radiofrequency ablation has been tested as a treatment option for bone metastases [8]. Currently, an off label use of Cryoablation techniques are being tested as another alternative for bone Mets palliation. The main goals of these treatments are improvement of quality of life and functional level. These goals can be further described:

1. Pain relief
2. Preservation and restoration of function
3. Local tumor control
4. Skeletal stabilization

Treatment with external beam radiation therapy (EBRT) is the standard of care for patients with localized bone pain, and results in the palliation of pain for many of these patients. Twenty to 30% of patients treated with radiation therapy do not experience pain relief [9-13]. Re-treatment rates are generally reported in the range of 10-25%. Many patients with relapsed pain or poor response to initial radiation may be lost to follow up or may not be referred back to oncologists for consideration of re-radiation. In addition to relapse and re-treatment, there is an increased risk of pathologic fracture in the peri-radiation period. The fracture rate reported in radiation studies is generally in the range of 1% to 8%. The hyperemic response weakens the adjacent bone and increases the risk of spontaneous fracture. Furthermore, patients who have recurrent pain at a site previously irradiated may not be eligible for further radiation therapy secondary to limitations in normal tissue tolerance. Hesitation on the part of physicians to use a larger dose may be related to increased long-term toxicity. Larger radiation dose produces a greater risk of complications such as fibrosis of normal soft tissue, which can cause a decrement in the quality of life in cases of life expectancy longer than 6 months. There may also be a greater incidence of acute side effects of nausea and vomiting if the treatment field includes the stomach. The percent of patients experiencing vomiting following EBRT ranges from about 5% to 30%.

A palliative treatment for painful bone metastases that is non-invasive, without long-term toxicity and having minimal complications would be a useful tool for treating physicians and also a beneficial option for patients suffering from painful bone metastases. Results of preliminary studies indicate that ExAblate treatment of painful bone metastases may be a beneficial treatment option [14, 15]. The ExAblate system is a non-invasive thermal ablation device used in the coagulation of various types of soft tissue. The ExAblate system has the potential to achieve the first three of the four previously mentioned goals in the treatment of bone tumors; namely pain relief, preservation and restoration of functional levels and local tumor control [11]. The ExAblate system used in the present study is a technological advance over the ExAblate 2000 fixed transducer system in terms of flexibility of use and reduction of positioning related pain to the patients. The ExAblate system used in this study conforms to the patient's body shape at the location of the bone mets location.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 and older
2. Patients who are able and willing to give consent and able to attend all study visits
3. Patients who are suffering from symptoms of bone metastases
4. One to 3 painful lesions.
5. Targeted tumor(s) are ExAblate device accessible and are located in ribs, extremities (excluding joints), pelvis, shoulders and in the posterior aspects of the following spinal vertebra: Lumbar vertebra (L3 - L5), Sacral vertebra (S1 - S5)
6. Patients with persistent distinguishable pain associated with up to 3 tumors of which a maximum of 2 tumors will be treated:

   o If patient has pain from additional sites that are not planned for treatment, the pain from the additional sites must be evaluated as being less intense by at least 2 points on the NRS compared to the site(s) to be treated.
7. Patient with NRS (0-10 scale) pain score ≥ 4 at the targeted tumors (i.e: both tumors targeted for treatment must have NRS ≥ 4) irrespective of medication
8. Targeted tumors (most painful) size up to 8 cm in diameter
9. Patient whose targeted (most painful) tumors are on bone and bone-lesion interface is deeper than 1cm from the skin.
10. Targeted (most painful) tumors clearly visible by non-contrast MRI, and ExAblate MRgFUS device accessible
11. Able to communicate sensations during the ExAblate MRgFUS treatment
12. At least 2 weeks since chemotherapy
13. No radiation therapy to targeted (most painful) tumors in the past two weeks

Exclusion Criteria:

1. Patients who either

   * Need surgical stabilization of the affected weight bearing bony structure (>7 fracture risk score, see Section 6.9) OR
   * Targeted tumor is at an impending fracture site of the weigh bearing bone (>7 on fracture risk score, see Section 6.9).

   OR

   o Patients with surgical stabilization of tumor site with metallic hardware
2. More than 3 painful lesions or more than 2 requiring immediate localized treatment
3. The targeted tumor(s) is (are) less than 2 points more painful compared to other non-targeted painful lesions on the site specific NRS.
4. Targeted tumor is in the skull
5. Patients on dialysis
6. Patients with life expectancy < 6-Months
7. Patients with an acute medical condition (e.g., pneumonia, sepsis) that is expected to hinder them from completing this study.
8. Patients with unstable cardiac status including:

   * Unstable angina pectoris on medication
   * Patients with documented myocardial infarction within six months of protocol entry
   * Congestive heart failure requiring medication (other than diuretic)
   * Patients on anti-arrhythmic drugs
9. Severe hypertension (diastolic BP > 100 on medication)
10. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
11. Patients with an active infection or severe hematological, neurological, or other uncontrolled disease.
12. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
13. KPS Score < 60 (See "Definitions" below)
14. Severe cerebrovascular disease (multiple CVA or CVA within 6 months)
15. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (can be up to 4 hrs of total table time.)
16. Target (most painful) tumor-bone interface is less then 1cm from nerve bundles, bowels or bladder.
17. Are participating or have participated in another clinical trial for the palliation of their targeted bone metastasis tumors in the last 30 days
18. Patients receiving chemotherapy or radiation (i.e., to the targeted lesion (s)) within the last two weeks
19. Patients unable to communicate with the investigator and staff.
20. Patients with persistent undistinguishable pain (pain source unidentifiable)
21. Targeted (most painful) tumors size > 8 cm in diameter
22. Targeted (most painful) tumors:

    * NOT visible by non-contrast MRI, OR
    * NOT accessible to ExAblate device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-09; Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Methodist Hospital Research Institute, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- See also: Sponsor's web page — http://www.insightec.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol was approved to treat 50 participants at up to six sites. The study was closed by the Sponsor after treating 17 participants at five sites.
Pre-assignment Details: Of the 37 subjects enrolled (signed consent), 11 subjects failed additional study requirements and 9 subjects exited the study prior to treatment. Seventeen subjects received the study Exablate treatment.
Period: Overall Study
Arm/Group | ExAblate 2100 Treatment
Started | 17
Completed | 14
Not Completed | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | ExAblate 2100 Treatment
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The baseline characteristics were tabulated for the treated subjects.
  Participants
    Hispanic | 3
    Black | 1
    White | 7
    Asian | 5
    Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Device Effects
Description: Adverse effects outcomes are reported in the adverse events module.
Time Frame: 3 months
Measure: Number; unit: Events
Arm/Group | ExAblate 2100 Treatment
Number analyzed (Participants) | 17
Events | 18

2. Secondary Outcome: Change in NRS Pain Scores From Baseline at 3 Months
Description: Efficacy was evaluated by change in Numerical Rating Scale (NRS) pain scores at 3 months post treatment The NRS is an 11 point scale (0-10) with 0 as no pain and 10 as the worst pain. Larger numbers in score change from baseline indicate improvement (decrease) in pain. Two points improvement has been reported as a clinically meaningful.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | ExAblate 2100 Treatment
Number analyzed (Participants) | 17
Score on a scale | 3.9 (1.1)

3. Secondary Outcome: Change Brief Pain Inventory - Pain Interference From Baseline at 3 Months
Description: Quality of life was evaluated using average change from baseline at 3 Months using the Pain Interference section of the Brief Pain Inventory (BPI-Pain Interference). Larger change from Baseline numbers indicate improved function. Pain Interference is the mean of seven questions scored on an 11-point scale of 0 (does not interfere) to 10 (completely interferes). A positive change from Baseline (higher values) at the 3 Month visit indicates improvement or a reduction in pain interference
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | ExAblate 2100 Treatment
Number analyzed (Participants) | 17
Score on a Scale | 3.3 (1.9)

ADVERSE EVENTS:
Time Frame: 3 Month
Arm/Group | ExAblate 2100 Treatment
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 4/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate 2100 Treatment (N=17)
Cancer Death (Hepatobiliary disorders) | 1 (1) — Subject died due to progression of Hodgkin's lymphoma with metastases.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate 2100 Treatment (N=17)
Sonication pain (Injury, poisoning and procedural complications) | 4 (6)
Post-procedure pain / discomfort (Injury, poisoning and procedural complications) | 3 (3)
Skin pain (no redness) (Injury, poisoning and procedural complications) | 1 (1)
Skin burn (Injury, poisoning and procedural complications) | 1 (1)
Bruise at injection site (Injury, poisoning and procedural complications) | 1 (1) — Related to IV catheter
Position pain (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Increased creatinine (Renal and urinary disorders) | 1 (1)
Post-procedure pain / discomfort (Injury, poisoning and procedural complications) | 1 (1) — Incidental to Device
Swelling (Injury, poisoning and procedural complications) | 1 (1)
Unanticipated Effects (Product Issues) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early leading to small numbers of subjects analyzed. The study was designed to enroll 50 subjects. Enrollment was terminated after enrolling 17 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No